CLINICAL TRIAL: NCT03709251
Title: High Intensity Walking to Reduce Frailty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 safety precautions and public health guidelines, the study was terminated early.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Margaret Danilovich, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00205686
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Walking (Experimental): HIW (70-80% Heart Rate max)
  Interventions: Behavioral: High Intensity Walking
- Casual Speed Walking (Experimental): Self selected pace
  Interventions: Behavioral: Casual Speed Walking

INTERVENTIONS:
Behavioral: High Intensity Walking — Intense walking activity at an intensity of 70-80% of the maximum heart rate
  Arms: High Intensity Walking
Behavioral: Casual Speed Walking — Moderate intensity (50-60% of Heart Rate maximum)
  Arms: Casual Speed Walking

SUMMARY:
The purpose of this study is to evaluate a physical therapist (PT) led gait training intervention for 100 older adults with pre-frailty or frailty. The goals of this study are To determine the effect of gait training intensity on frailty, mobility, physical functioning, and quality of life, as well as balance and healthcare utilization.

DETAILED DESCRIPTION:
Frailty is a leading cause of dependency among older adults, affects up to 60% of older adults, and is associated with an increased risk for falls, hospitalizations, institutionalization, and death. Exercise is the most widely recommended treatment for improving physical function among the frailty, but the optimal type or intensity of exercise is unknown. Walking is a preferred physical activity among older adults, however, there are no clear guidelines on the best intensity of walking to reduce frailty. The specific goal of this project is to compare a high intensity walking (HIW) intervention (70-80% of heart rate maximum) to a moderate intensity walking (MIW) intervention (50-60% of heart rate maximum) for pre-frail or frail older adults to determine the impact on frailty, mobility, balance, quality of life, and healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

* Receiving services from CJE SeniorLife
* Pre-frailty or frailty as determined on the SHARE-FI.
* Able to ambulate at least 10 feet with moderate assistance (<50% physical assistance) or less. Participants will be able to use their assistive device (e.g. cane or walker) during sessions.
* > 65 years of age
* Provision of informed consent and clearance for participation as determined by the Exercise and Screening for You (EASY)

Exclusion Criteria:

* Uncontrolled cardiovascular, metabolic, renal, or respiratory disease that limits exercise participation (e.g., previous heart attack within 3 months of enrollment or uncontrolled diabetes)
* Resting blood pressure > 180/110 mmHg.59

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Change in frailty as measured by the Survey of Health, Ageing, and Retirement in Europe-Frailty Instrument (SHARE-FI) | Baseline, Week 9, Month 6
  Survey of Health, Ageing, and Retirement in Europe-Frailty Instrument (SHARE-FI) which assesses fatigue, appetite, weakness, walking difficulties, and low physical activity

SECONDARY OUTCOMES:
Improved mobility as measured by gait speed | Baseline, Week 9, Month 6
  Measures related to overall health and mobility
Improved mobility as measured by 6 Minute Walk Test | Baseline, Week 9, Month 6
  Measures related to mobility
Improved mobility as measured by Time Up and Go | Baseline, Week 9, Month 6
  Measures related to mobility
Improved physical function on the Short Physical Performance Battery | Baseline, Week 9, Month 6
  Provide an overall assessment of functional status and physical performance
Improved balance as measured by the Berg Balance Scale | Baseline, Week 9, Month 6
  The Berg Balance Scale is a valid and reliable 14 item tool to evaluate static and dynamic balance among older adults. Minimum Score 0 to Maximum Score 56. • Score of < 45 indicates individuals may be at greater risk of falling
Monthly self reports of Health Care Utilization | Baseline, Week 9, Month 3, Month 4, Month 5, Month 6
  Monthly self-reports of number of falls, number of hospitalizations, and number of emergency room visits
Patient Reported Outcomes Measure Information System (PROMIS) Global Health | Baseline, Week 9, Month 6
  assess subjective measures of physical and mental health, pain, and quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Univiersity Department of Physical Therapy and Human Movement Sciences, Chicago, Illinois, United States